CLINICAL TRIAL: NCT04732858
Title: Educational Interventions to Integrate Surgical Staff Within Medical Units During the COVID-19 Pandemic: EDUCOVID Cross-sectional, E-survey
Brief Title: Educational Interventions for Surgeons During COVID-19 Pandemic: Cross-sectional, E-survey
Acronym: EDUCOVID
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP201297
Record Dates: First submitted 2021-01-29; First posted 2021-02-01 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2020-11

CONDITIONS: COVID-19
Keywords: 2019-nCoV; COVID-19; Pandemic; Educational intervention; Medical education
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cross sectional e-Survey on surgeons exposed to any educational intervention — Educational intervention was considered as any procedure or program to facilitate the acquisition of basic skills about the disease, its ramifications and treatment2,6,7:
  * Education in infectious disease, including
    * "pandemic" training for health personnel
    * Personal protective equipment (PPE) and protection.
    * Specific speed-training focusing on environmental control (decontamination area, dressing...), personal protection, hand hygiene, sample management, risky gestures, control measures.
  * Intensive care education:
    * mechanical ventilation
    * airways management
    * emergencies and cardiovascular drugs
    * Intensive care monitoring systems
  * Basic nurse skills
  * COVID-specific clinical management

SUMMARY:
The coronavirus disease 2019 (COVID-19) pandemic required a rapid surge of healthcare capacity to face a growing number of critically ill patients. For this reason, a support reserve of physicians, including surgeons, were required to be reassigned to offer support. Given the time shortage for trainers and trainees, time and cost-efficient programs to gain maximal benefit from short rotations for several physicians at one time are required 8. In case of pandemics, blending face-to-face education to e-learning seems sustainable, with online resources being scalable and more cost effective than other methods 9.

DETAILED DESCRIPTION:
The aim of this study was to realize a survey on the educational programs (hospital based or web-based), during the COVID-19 pandemic, and their impact on behavior change, satisfaction and knowledge of the target population of surgeons.

ELIGIBILITY:
Inclusion Criteria:

* residents, fellows, consultants and physicians of any grade and affiliated to any surgical specialty

Exclusion Criteria:

* Mecical speciality

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This survey was conceived as open to residents, fellows, consultants and physicians of any grade and affiliated to any surgical specialty.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Kirkpatrick level 3 on a 5-modalities Likert scale | once at the time of survey
  The primary endpoint of the e-survey was to explore the effectiveness of educational interventions experienced by responders, considered as a whole "bundle" (and not one-by-one), among the surgeons exposed to a training program, on behavior change (Kirkpatrick level 3) in their daily role during their re-affectation within a medical COVID-unit. Behavior change represents a change in the daily role of healthcare professionals (for example, referral of patients with suspected COVID to the most appropriate screening and care pathway). For this survey, we considered subjective measures (self-assessment on a Likert scale on 5 modalities) of behavior change.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaele BRUSTIA, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Assistance Publique Hôpitaux de Paris - GHU AP-HP Hôpitaux Universitaires Henri-Mondor, Créteil, France